CLINICAL TRIAL: NCT02181881
Title: Relationship Factors and HIV Treatment Adherence
Brief Title: DuoPACT Pilot Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: R01NR010187 (NIH); R01NR010187 (NIH)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DuoPACT (Active Comparator): A 6-session HIV medication adherence support program for couples.
  Interventions: Behavioral: DuoPACT
- Life Steps (Active Comparator): A 3-session HIV medication adherence support program for individuals.
  Interventions: Behavioral: Life Steps
- Treatment as usual (TAU) (No Intervention): HIV positive individuals will continue to follow their current HIV treatment plan.

INTERVENTIONS:
Behavioral: DuoPACT — Intervention sessions are administered weekly by a counselor.
  Arms: DuoPACT
Behavioral: Life Steps — Intervention sessions are administered weekly by a counselor.
  Arms: Life Steps

SUMMARY:
The investigators will pilot test the intervention by randomizing 30 couples to one of three conditions: 1) DuoPACT, the newly-developed couples intervention; 2) Life Steps, a standardized antiretroviral adherence intervention for HIV+ individuals; and 3) a treatment as usual (TAU) assessment-only control condition. After randomization, intervention sessions will be delivered weekly (6 DuoPACT sessions, or 3 Life Steps sessions). All couples will be assessed pre/post intervention to evaluate intervention acceptability and feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. Gay male couple.
2. One or both partners must be HIV positive and on antiretroviral medications.

Exclusion Criteria:

Must be able to consent to and follow study protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the intervention | 3 months
  All participants are assessed post intervention to evaluate intervention satisfaction and acceptability.

SECONDARY OUTCOMES:
Feasibility | 3 months
  All participants are assessed post intervention to evaluate the study's feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Mallory O Johnson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Center for AIDS Prevention Studies, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No